CLINICAL TRIAL: NCT04103554
Title: A Multicenter, Randomized, Open-label, Parallel Group, Pilot Study to Evaluate the Use of Sacubitril/Valsartan in HeartMate 3 LVAD Recipients
Brief Title: Sacubitril/Valsartan in Left Ventricular Assist Device Recipients
Acronym: ENVAD-HF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Maja Cikes, Associate professor, MD, PhD, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENVAD-HF
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
Keywords: LVAD (Left Ventricular Assist Device); sacubitril/valsartan; heart failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sacubitril/valsartan (Experimental)
  Interventions: Drug: Sacubitril-Valsartan
- Standard of care (Active Comparator): Standard of care for treating blood pressure per center protocols
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Sacubitril-Valsartan 24/26 mg BID, 49/51 mg BID, 97/103 mg BID
  Arms: sacubitril/valsartan
Drug: Standard of care — standard of care used for treating BP
  Arms: Standard of care

SUMMARY:
The primary objective of this prospective randomised study is to assess the safety and tolerability of sacubitril/valsartan compared with standard of care used for treating BP in patients that have been implanted with the Heart Mate 3 LVAD (events of special interest - all cause death, right ventricular failure, bleeding events, deterioration in renal function, hyperkalemia, symptomatic hypotension).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. ≥18 years of age, male or female
3. Recently implanted HeartMate 3 LVAD recipients, in stable condition and deemed ready for discharge or chronic, stable, ambulatory HeartMate 3 LVAD carriers implanted within 1 year prior to enrolment

1. Current acute decompensated HF (including right ventricular failure) requiring therapy with intravenous diuretics or vasodilators and/or inotropic drugs within the past 48 hours 2. History of hypersensitivity to sacubitril/valsartan or to drugs of similar chemical classes, patients with a known history of angioedema 3. Patients with mean blood pressure ≤75 mmHg (systolic blood pressure i.e. Doppler opening blood pressure ≤90 mmHg in those pulsatile and measured by Doppler method) or symptomatic hypotension 4. eGFR < 30 mL/min/1.73m2 as calculated by the Modification in Diet in Renal Disease (MDRD) formula at Visit 1 5. Patients with serum potassium >5.4 mmol/L (mEq/L) at Visit 1 6. Hemodynamically unstable patients or those with ongoing MCS other than LVAD or those with planned biventricular support 7. Hemodynamically significant aortic insufficiency in the opinion of the investigator 8. Irreversible end-organ dysfunction 9. Previous sacubitril/valsartan use while on LVAD support 10. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or other major CV surgery, percutaneous coronary intervention (PCI) or carotid angioplasty within 30 days prior to enrolment 11. Life-threatening or uncontrolled dysrhythmia, including symptomatic or sustained ventricular tachycardia and atrial fibrillation or flutter with a resting ventricular rate >110 bpm at enrolment 12. Any surgical or medical condition, which in the opinion of the Investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study 13. Active infection with hemodynamic compromise 14. hemoglobin (Hgb) <8 g/dl 15. body mass index (BMI) > 45 kg/m2 16. Congenital heart disease 17. Coronary or carotid artery disease or valvular heart disease likely to require surgical or percutaneous intervention within the 6 months after enrolment 18. Evidence of hepatic disease as determined by any one of the following: SGOT (AST) or SGPT (ALT) values exceeding 3x ULN, bilirubin >1.5 mg/dl at Visit 1 19. Pregnant or nursing (lactating) women and women of child-bearing potential unless they are using highly effective methods of contraception

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Freedom from all-cause death, deterioration in renal function (reaching end-stage renal disease (ESRD), renal death or 50% decline in eGFR), hyperkalemia or symptomatic hypotension | 3 months
  * End-stage renal disease defined as one of the following:
    1. Initiation of dialysis (e.g., hemodialysis, peritoneal dialysis, or continuous venovenous hemodialysis), continuing for ≥ 20 days without known recovery of renal function
    2. Initiation of dialysis with death before 30 days (excludes dialysis events associated with acute kidney injury with death before 30 days)
    3. A drop in eGFR from baseline (randomization, i.e. Visit 101) to a value <15 mL/min/1.73m2 on two consecutive measurements separated by≥ 20 days
    4. Occurrence of kidney transplantation
  * 50% sustained decline in eGFR: 50% decline from baseline (Randomization, Visit 101) as determined by 2 consecutive post-baseline measurements separated by ≥ 20 days
  * Hyperkalemia: serum potassium ≥6.0 mmol/L [mEq/L]) Hypotension: symptomatic reduction in blood pressure requiring withdrawal of study medication or any BP lowering medication

SECONDARY OUTCOMES:
Change in NT-proBNP from enrolment to 8 weeks | 8 weeks
Change in Burden of hemocompatibility (hemocompatibility score) | 3 months, 12 months
Number of RV failure events | 3 months, 12 months
Time to first unplanned hospitalisation | 3 months, 12 months
Number of unplanned hospitalizations | 3 months, 12 months
Change in blood-pressure lowering medications | 3 months, 12 months
Change in eGFR values | 3 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maja Cikes, MD, PhD, Principal Investigator — University of Zagreb School of Medicine
Locations (6):
- Croatia (2):
  - University Hospital Centre Zagreb, Zagreb
  - University Hospital Dubrava, Zagreb
- IKEM, Prague, Czechia
- Netherlands (2):
  - Erasmus Medical Centre, Rotterdam
  - University Medical Centre Utrecht, Utrecht
- John Paul II Hospital, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided